CLINICAL TRIAL: NCT06713109
Title: Motivasyonel Görüşme Il Verilen Emzirme Danışmanlığının Emzirme Sorunu Ve Kaygıya Etkisi
Brief Title: The Effect of Breastfeeding Counselling with Motivational Inter-viewing Technique on Breastfeeding Problems and Anxiety
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: semiha izgordu (Other)
Collaborators: Marmara University (Other)
Responsible Party: Sponsor-Investigator, semiha izgordu, Midwife, Uskudar University
Organization: Uskudar University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 6135142-020-143
Record Dates: First submitted 2024-11-07; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Breast Feeding; Anxiety; Motivational Interviews
Keywords: breastfeeding; motivational interviewing; anxiety
MeSH Terms: conditions — Breast Feeding; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: breastfeeding problems anxiety motivational interviewing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- arm1 (No Intervention): Will receive standard breastfeeding training and after 3 weeks the final test will be administered
- arm2 (Experimental): A motivational interview will be conducted to get information about the breastfeeding problem and the level of loss and to try to support it with interviews.
  Interventions: Behavioral: Motivational interview techniques

INTERVENTIONS:
Behavioral: Motivational interview techniques — Motivational interviews will be conducted 4 times. As a result of these interviews, the breastfeeding problem or anxiety in the mother will be evaluated and the effectiveness of the interview will be solved.
  Arms: arm2

SUMMARY:
The primary aim of this study was to investigate the effect of motivational interviewing technique on breastfeeding problems and loss.

H1:The breastfeeding problems score of the mothers who received motivational interviewing was lower than the mothers who received standard care.

H 2: The anxiety level score of mothers who received motivational interviewing is lower than that of mothers who received standard care.

H3: The rate of exclusive breastfeeding of mothers who received motivational interviewing is higher than that of mothers who received standard care.

DETAILED DESCRIPTION:
The data elements to be used in the study are as follows:

'Personal Information Form (Appendix-1)', "Breastfeeding Problems Assessment Scale (Appendix-2)" to determine the problems experienced by mothers regarding breastfeeding, and "State Anxiety Scale (Appendix-3)" to determine the anxiety level of mothers will be used to collect the data. 'Informed Consent Form (Appendix-4)' will be filled in and permission to participate in the study will be obtained.

Appendix 1- Personal Information Form A personal information form was prepared by reviewing the literature (Gölbaşı et al.) The information form questioning the socio-demographic, obstetric and breastfeeding characteristics of the mothers was prepared by the researcher and consisted of 19 items in total.

Appendix-2 Breastfeeding Problems Assessment Scale (BPSAS) Originally named 'Breastfeeding Experience Scale', the ESBS was developed by Karen Wambach in 1990 to evaluate mothers' breastfeeding experiences . The Turkish validity and reliability of the scale was conducted in 2019 . The original scale has a 5-point Likert type and consists of 5 sub-dimensions and 30 items. The scale consists of two parts. The first part consists of 18 items and evaluates breastfeeding problems. The second part consists of items 19-30 and assesses mothers' weaning experiences and formula supplementation practices. The Turkish version of the scale includes only the first part and consists of 18 items and 5 sub-dimensions. The 5 sub-dimensions of the scale (mechanical concerns; 16, 6, 4, 11, 14, process concerns; 12, 9, 8, 5, 3, milk insufficiency concerns; 13, 15, 10, breast concerns; 2, 1, 7, social concerns; 18, 17) were determined by confirmatory factor analysis. Scale items are graded as 1; not at all, 2; mild, 3; moderate, 4; severe, 5; unbearable. Each item is scored between 1 and 5. The minimum and maximum scores that can be obtained from the scale are 18-90. High scores obtained from the scale indicate that breastfeeding problems are severe. Cronbach's alpha coefficient for the evaluation of the reliability of the 18 items in the Breastfeeding Problems Assessment Scale was found to be 0.776. Cronbach's alpha values of the scale sub-dimensions; mechanical concerns; 0.852, process concerns; 0.712, milk insufficiency concerns; 0.766, breast concerns; 0.748, social concerns; 0.789 were found. It was found that there was no difference between the test-retest measurements of the scale and its invariance over time was determined. It was determined that the Breastfeeding Problems Assessment Scale is an appropriate measurement tool for assessing the problems of breastfeeding mothers in Turkish society.

Appendix 3- State Anxiety Inventory (STAI State Anxiety Inventory) State Anxiety Scale is a self-assessment questionnaire consisting of short statements. The State Anxiety Scale requires the individual to describe how he/she feels at a certain moment and under certain conditions and to answer by taking into account his/her feelings about the situation he/she is in. It consists of 20 questions in total.

The feelings or behaviours expressed in the items of the state anxiety scale consist of 1) not at all, 2) a little, 3) a lot and 4) completely according to the severity of the experience. Developed in 1964 by Spielber-ger and Gorsuch, the inventory aims to measure trait and state anxiety levels in normal and non-normal individuals.

After the adaptation and standardisation of the scale into Turkish by Öner and Le Compte in 1974-1977, the inventory was used in studies involving Turkish youth and adult groups.

There are two types of statements in the scale. These can be called (1) direct or straight statements and (2) re-verse statements. Direct statements express negative emotions, whereas reversed statements express positive emotions. When scoring these second type of statements, those with a weight value of 1 are converted to 4 and those with a weight value of 4 are converted to 1. In direct statements, answers with a value of 4 indicate that anxiety is high. In inverted statements, answers with a value of 1 indicate high anxiety and answers with a value of 4 indicate low anxiety. The expression 'I am restless' can be shown as an example of direct statements and the expression 'I feel calm' can be shown as an example of inverted statements. In this case, if an option with a weight of 4 is selected for the expression 'I feel restless' and an option with a weight of 1 is selected for the expression 'I feel calm', these answers reflect high anxiety. There are ten inverted statements in the state anxiety scale. These are items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20.

In the reversed statements, the ones with a value of 1 turn into 4, and the ones with a value of 4 turn into 1 and scoring is done. The score obtained in the total of both scales takes minimum 20 and maximum 80 values. A high total score indicates an increase in anxiety level, while a low score indicates a decrease in anxiety level . A total score above 60 points indicates that the individual needs professional support.

0-40 points: No anxiety 41-60 points: Mild anxiety 61>points: Severe anxiety. Annex-4 Informed Consent Form The consent form was prepared by the researcher and the consent of the intervention and control groups will be obtained separately.

ELIGIBILITY:
Inclusion Criteria:

* Having a healthy 1-3 month old baby
* Being identified as having a breastfeeding problem
* To be at least primary school graduate
* To be able to communicate by telephone
* To come to the Family Health Centre for motivational talks

Exclusion Criteria:

* Having a baby with anomalies
* Having a baby younger than 1 month and older than 3 months
* Having a medical illness that prevents breastfeeding
* Communication problems
* Not accepting motivational interviewing
* The presence of any psychiatric illness

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Nursing mothers with a 1-month-old baby
Enrollment: 64 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-27 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
The effect of motivational interviewing on breastfeeding | three weeks from the start of the interview
  Breastfeeding Problems Assessment Scale and State Anxiety Inventory scores will be collected and statistical analysis will be performed by spss software and expert statistician opinion will be obtained.
The effect of motivational interviewing on anxiety | three weeks from the start of the interview
  Breastfeeding Problems Assessment Scale and State Anxiety Inventory scores will be collected and statistical analysis will be performed by spss software and expert statistician opinion will be obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara Üniversitesi Pendik Eğitim Aile Sağlığı Merkezi, Istanbul, tuzla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
kimlerle paylaşılacağından emin değilim